CLINICAL TRIAL: NCT01223170
Title: eRehab: Can Information and Communication Technology (ICT) Enhance Self-management of Cardiovascular Disease?
Acronym: eRehab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of North Norway (Other)
Collaborators: Helse Nord (Industry); LHL Helse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UNN-NST-eRehab-01
Record Dates: First submitted 2010-09-06; First posted 2010-10-18 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Cardiovascular Diseases
Keywords: Tailoring; Cardiac rehabilitation; Internet based intervention; Exercise; Cardiovascular Disease rehabilitation
MeSH Terms: conditions — Cardiovascular Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Internet-based intervention (Experimental): Behavioral: Tailored content Behavioral: Generic Internet-based information Behavioral: Discussion forum Behavioral: Behavioral monitoring
  Interventions: Behavioral: Tailored content; Behavioral: Generic Internet-based information; Behavioral: Discussion forum; Behavioral: Behavioral monitoring
- Control (Placebo Comparator): Behavioral: Generic Internet-based information Behavioral: Discussion forum
  Interventions: Behavioral: Generic Internet-based information; Behavioral: Discussion forum

INTERVENTIONS:
Behavioral: Tailored content — Participants will have access to content tailored for Stage of Change, Regulatory Focus and Self-Efficacy.
  Other Names: Internet based intervention
  Arms: Enhanced Internet-based intervention
Behavioral: Generic Internet-based information — Access to a website with general information about Cardiovascular Disease and self-management, including diet, physical activity, smoking and medications.
  Other Names: Internet based intervention
Behavioral: Discussion forum — Access to a discussion forum for Cardiovascular Disease Rehabilitation.
  Other Names: Internet based intervention
Behavioral: Behavioral monitoring — Participants will be offered behavioral monitoring, based on data collected from online self-reports and from activity sensors built into mobile phones.
  Other Names: Internet based intervention
  Arms: Enhanced Internet-based intervention

SUMMARY:
Cardiovascular Diseases (CVD) according to the World Health Organization (WHO) are leading causes of death and represent 30% of all global deaths and 48% of the deaths in Europe. Moreover, the current trends predict increase in deaths caused by Cardiovascular Diseases over the next years. Secondary preventive efforts can decrease mortality risk as well as improve health among Cardiovascular Disease patients.

This study suggests an innovative approach in supporting the self-management of Cardiovascular Disease patients after rehabilitation. The implied Randomized Controlled Trial has two arms and aims to investigate the effectiveness of tailoring in an Information and Communication Technology (ICT) based intervention. The tailoring will be based on concepts derived from health psychology theories, and will contribute in their further development. More specifically:

* Aim 1: To assess the needs of CVD rehabilitation patients that can potentially be met through the use of ICT.
* Aim 2: To assess the effects of a tailored Internet-based intervention on maintenance of self-management behaviors after a rehabilitation stay. Hypothesis: The intervention group (tailored) will have higher adherence a) to the Internet-based intervention, and b) to self-management.
* Aim 3: To assess the effect of mobile technology with activity sensors on physical activity. Hypothesis: There will be a relationship between the data collected from activity sensors and the self-reported physical activity levels.

DETAILED DESCRIPTION:
A parallel group, cluster randomized controlled trial. The study population is adult participants of a cardiac rehabilitation programme in Norway with home Internet access and mobile phone, who in monthly clusters are randomized to the control or the intervention condition. Participants have access to a website with information regarding cardiac rehabilitation, an online discussion forum and an online activity calendar. Those randomized to the intervention condition, receive in addition tailored content based on models of health behaviour, through the website and mobile text messages. The objective is to assess the effect of the intervention on maintenance of self-management behaviours after the rehabilitation stay. Main outcome is the level of physical activity one month, three months and one year after the end of the cardiac rehabilitation programme. The randomization of clusters is based on a true random number online service, and participants, investigators and outcome assessor are blinded to the condition of the clusters.

The study suggests a theory-based intervention that combines models of health behaviour in an innovative way, in order to tailor the delivered content. The users have been actively involved in its design, and because of the use of Open-Source software, the intervention can easily and at low-cost be reproduced and expanded by others. Challenges are the recruitment in the elderly population and the possible underrepresentation of women in the study sample

ELIGIBILITY:
Inclusion Criteria:

* History of cardiovascular disease
* Admission to the collaborating rehabilitation center

Exclusion Criteria:

* Technological illiteracy
* Inability to access internet at home

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Duration and Intensity of Physical Activity | 1 month, 3 months and 12 months after discharge

SECONDARY OUTCOMES:
Use of online intervention | 1 month after discharge
Use of online intervention | 3 months after discharge
Use of online intervention | 12 months after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Silje Camilla Wangberg, PhD, Principal Investigator — Kompetansesenter for Rus, Nord-Norge
Locations (1):
- Skibotn Rehabilitering, Ivgobahta, Troms, Norway

REFERENCES:
- [Background] Antypas K, Wangberg SC. E-Rehabilitation - an Internet and mobile phone based tailored intervention to enhance self-management of cardiovascular disease: study protocol for a randomized controlled trial. BMC Cardiovasc Disord. 2012 Jul 9;12:50. doi: 10.1186/1471-2261-12-50. PMID 22776554
- [Result] Antypas K, Wangberg SC. An Internet- and mobile-based tailored intervention to enhance maintenance of physical activity after cardiac rehabilitation: short-term results of a randomized controlled trial. J Med Internet Res. 2014 Mar 11;16(3):e77. doi: 10.2196/jmir.3132. PMID 24618349
- [Derived] Antypas K, Wangberg SC. Combining users' needs with health behavior models in designing an internet- and mobile-based intervention for physical activity in cardiac rehabilitation. JMIR Res Protoc. 2014 Jan 10;3(1):e4. doi: 10.2196/resprot.2725. PMID 24413185
- See also: Norwegian Centre for Integrated Care and Telemedicine — http://www.telemed.no